CLINICAL TRIAL: NCT07212478
Title: Comparison Between Pelvic Floor Muscle Training and Pilates Exercises for Postmenopausal Women With Urinary Incontinence
Brief Title: Pelvic Floor Muscle Training vs. Pilates Exercises for Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Laís Campos de Oliveira, Doctor Teacher Laís Campos de Oliveira, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5.264.703
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Urinary Incontinence , Stress
Keywords: Post-menopause; Pilates; Muscle training of pelvic floor
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: The interventions will last twelve weeks, twice a week, for one hour, on alternating days.
  1. The pelvic floor muscle training group protocol will consist of four sets of ten maximal contractions, held for at least six seconds, followed by five rapid contractions at the end of each set. Each set will be performed in a different position: first lying on your side, second sitting, third on all fours, and fourth standing.
  2. The Pilates exercise group protocol will consist of 10 exercises, four specific to stretching and six for muscle strengthening.
Who Masked: Outcomes Assessor
Masking Description: The randomization of the sample will be confidential. A professional in the field who is unaware of the study and the participants will perform the draw through random numbers that will distribute the participants into two groups: Pelvic Floor Muscle Training Group (TMAP) (n= 12) and Pilates Exercise Group (PE) (n= 12). This same professional will deliver the answers in opaque envelopes, which will be sealed and contain the answer. Participants will be duly informed that they can be allocated to either of the two groups at the time of recruitment and selection and, in addition, the participants and the responsible researchers will know in which group each woman will participate at the time of delivery of the envelopes. The evaluations will be carried out before and after three months of interventions, by the same professionals, experienced in these evaluations, who will be blind to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Training (Active Comparator): Active Comparator: Pelvic floor muscle training (PFMT) For the intervention of the PFMT group, which is noninvasive, a physical therapist experienced in this type of training will carry out the sessions, which will be individualized, in a specific room for care ocused on pelvic physiotherapy, with a stretcher, air conditioning and a lock on the door, for the patient to feel safe.
  Interventions: Other: PFMT
- Pilates exercises (PE) (Experimental): For the Pilates group intervention, in the first week, the protocol will be used to familiarize participants with the exercises, demonstrating the correct execution of the movements and explaining each principle of the method: concentration, centering, precision, breathing, control, and fluidity. Ten Pilates mat exercises will be performed: 1- Rolling; 2- Swan; 3- Forward Leg Pull; 4- Bridge; 5- Hundred; 6- Crossover; 7-Wall Slide; 8- Side Kick: Inner Thigh Raise; 9- Arms Forward; 10- Forward Spine Stretch.
  Interventions: Other: Pilates exercises

INTERVENTIONS:
Other: PFMT — O PFMT consistirá em 10 contrações voluntárias máximas que devem ser mantidas por pelo menos 6 segundos. Os participantes serão incentivados a sustentar a contração máxima por um tempo maior a cada semana. O intervalo entre as contrações será de segundos. Os participantes realizarão 4 séries de 10 contrações e, ao final de cada série de 10 contrações, serão realizadas cinco contrações rápidas. Cada série será realizada em uma posição: deitado em decúbito lateral; sentado; de quatro apoios e em pé.
  Arms: Pelvic Floor Muscle Training
Other: Pilates exercises — The Pilates group will perform 10 solo exercises, containing stretching and strengthening for the main muscle groups, with a single series of 10 repetitions.
  Arms: Pilates exercises (PE)

SUMMARY:
Urinary incontinence (UI) affects approximately 40% of postmenopausal women and is therefore considered a public health problem. Conservative treatment is recommended, and pelvic floor muscle training (PFMT) is considered the gold standard for this condition.

However, other exercise options have been studied, such as Pilates exercises, which focus on stabilizing muscles and require voluntary contraction of the pelvic floor muscles. The literature remains inconclusive regarding the effects of Pilates exercises on urinary incontinence and pelvic floor muscle function. Objective: To compare the effects of 3 months of muscle training, through PFMT and Pilates exercises, on improving UI in postmenopausal women. Methods: Twenty-four postmenopausal women with urinary incontinence will be randomized into two intervention groups: pelvic floor muscle training and mat Pilates exercises. Assessments will be conducted before and after three months of intervention and will include the following instruments: urinary incontinence and quality of life, assessed using the International Consultation of Urinary Incontinence Short Form (ICIQ-UI-SF) questionnaire; a 7-day voiding diary to identify potential modifiable factors related to urination and its frequency; a Pad test to identify and quantify UI; the Female Sexual Function Index to assess female sexual function; and pelvic floor muscle strength and endurance by bidigital palpation using the PERFECT test. Shapiro-Wilk tests will be used to assess normality, Student's t-test or Mann-Whitney U test according to parametric or nonparametric distribution, and ANCOVA will be used to compare groups post-intervention, considering a 95% confidence interval (p<0.05). Data will be processed using SPSS 25.0.

DETAILED DESCRIPTION:
The sample will consist of 24 postmenopausal women, that is, who have not menstruated for at least one year and are between 50 and 70 years of age. The sample size was determined by a sample calculation performed in the Bioestat 5.3 program (Mamirauá Institute, Amazonas, Brazil), taking into account the values of the ICIQ_SF (International Consultation on Incontinence Questionnaire - Short Form) instrument, made available in a previous study (SCHRADER et al., 2017). In this case, the post-intervention mean and standard deviation between the Pilates (8.71 ± 2.98) and PFMT (5.14 ± 2.73) groups were used, with the test power at 80% and an alpha value of 0.05, which generated the need for 10 participants in each group. To account for potential sample losses, 15% of participants were added to each of the two groups, totaling 12 women in each group.

Descriptive data analysis will be expressed as mean, standard deviation, and delta percentage difference. Normality will be verified using the Shapiro-Wilk test. To assess for differences between groups regarding baseline characteristics (age, weight, height, and BMI) at the pre-intervention stage, the Student's t-test for independent samples or the Mann-Whitney U test will be used if the data present a parametric or nonparametric distribution, respectively. For comparison between groups post-intervention, ANCOVA will be used, with baseline data used as covariates. If the data present nonparametric characteristics, the comparison between groups will be made using the Mann-Whitney U test, considering the difference between pre- and post-intervention. The accepted confidence interval will be 95% (p<0.05). Data will be processed using SPSS 25.0. Effect sizes (Cohen's d) will be calculated and considered small (0.20), medium (0.50), or large (0.80). For effect size calculations, the GPower 3.1 program (Franz Faul, Universitat Kiel, Germany) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being naturally post-menopause (at least one year without menstruating);
* Demonstrate independence to carry out activities of daily living;
* Have a report of urinary loss when performing physical exertion.

Exclusion Criteria:

* Women who have had hysterectomy or oophorectomy surgery;
* Women who underwent cancer treatment with hormone therapy;
* Present cognitive deficits or neurological diseases;
* Practice any type of physical activity regularly in the last six months; Present inability to hire PFM (Oxford Scale < 1);
* Report pain or discomfort in the vulva or vagina;
* Present dyspareunia, vaginismus or pelvic organ prolapse greater than grade II in the Baden-Walker classification;
* Present symptoms of urinary infection at the time of evaluation;
* Have participated in previous pelvic floor reeducation programs.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Voiding diary | 12 weeks
  Identifies the frequency of urinary leakage. The participant will record, over the course of 7 days, at home, the number of episodes of urinary leakage during some effort, such as coughing, sneezing or jumping. If there are more than 3 urinary losses within a 7-day interval, the test is positive for UI.
International Consultation of Urinary questionnaire Incontinence Short Form (ICIQ-UI-SF) | 12 weeks
  Specific quality of life questionnaire for each aspect related to UI. It consists of four questions; the sum of the first three questions gives the score, and the fourth describes the type of UI. The maximum total score is 21, and the higher the score, the worse the UI severity and disorder.
PERFECT test | 12 weeks
  As a complement to the manometric evaluation, bidigital palpation will be performed. The PFM strength and resistance level will be classified using the modified Oxford scale, where 0 is the absence of muscle strength and 5 means a strong contraction with movement correct "squeeze" and "suction". Participants will attempt maximum contractions in terms of strength and endurance three times, with 30-second rest intervals between contractions. The closer to a score of 5, the better the MAP.
FSFI Questionnaire (Female Sexual Function Index) | 12 weeks
  To assess women's sexual function, the domains: desire, arousal, lubrication, orgasm, satisfaction and pain are used. It has 19 items. Each question presents a possibility of response with a pattern from 0 to 5, where at the end you can have the result of the scores of each domain and also of the total score, where values below or equal to 26.55 indicate sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Laís Campos de Oliveira, PhD, Principal Investigator — Universidade Estadual do Norte do Paraná
Locations (1):
- Laís Campos de Oliveira, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No